CLINICAL TRIAL: NCT03946514
Title: Efficacy and Safety of a Single-pill Fixed Combination of Sufficient Losartan/Hydrochlorothiazide in Chinese Hypertensive Patients (FOCUS)
Brief Title: Efficacy and Safety of a Single-pill Fixed Combination of Sufficient Losartan/Hydrochlorothiazide in Chinese Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOCUS
Record Dates: First submitted 2019-05-05; First posted 2019-05-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
Keywords: Blood pressure; single-pill fixed combination; losartan/hydrochlorothiazide; amlodipine/hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly divided into two groups, taking losartan 100 mg/hydrochlorothiazide 25 mg fixed combination once a day or amlodipine besylate tablets (5 mg/tablet) + hydrochlorothiazide tablets (25 mg/tablet) once a day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan/hydrochlorothiazide group (Experimental)
  Interventions: Drug: losartan/hydrochlorothiazide
- amlodipine/hydrochlorothiazide group (Active Comparator)
  Interventions: Drug: amlodipine/hydrochlorothiazide

INTERVENTIONS:
Drug: losartan/hydrochlorothiazide — losartan 100 mg/hydrochlorothiazide 25 mg single-pill combination
  Arms: losartan/hydrochlorothiazide group
Drug: amlodipine/hydrochlorothiazide — amlodipine besylate tablets (5 mg / tablet) + hydrochlorothiazide tablets (25 mg / tablet)
  Arms: amlodipine/hydrochlorothiazide group

SUMMARY:
1. Study name: Efficacy and safety of a single-pill fixed combination of sufficient losartan/hydrochlorothiazide in Chinese hypertensive patients (FOCUS)
2. Medicine: Losartan 100 mg/hydrochlorothiazide 25 mg single-pill fixed combination; amlodipine besylate tablet (5 mg/tablet); hydrochlorothiazide tablets (25 mg/tablet)
3. Rationale: Angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) combined with thiazide diuretic (DIU), which is the preferred combination for most hypertension guidelines. However, the efficacy and safety of losartan 100 mg/hydrochlorothiazide 25 mg single-pill fixed combination evaluated by ambulatory blood pressure are still lack of clinical evidence.
4. Objective: To evaluate the efficacy and safety of losartan 100 mg/hydrochlorothiazide 25 mg fixed combination for ambulatory blood pressure after 8 weeks therapy in patients over 18 years with grade 1 or 2 hypertension either newly diagnosed or with blood pressure not controlled with monotherapy.
5. Study design: This study is a multi-center, randomized and controlled clinical trial with two equally sized treatment groups: losartan/hydrochlorothiazide single-pill fixed combination and amlodipine/hydrochlorothiazide.
6. Study population: Men and Women aged over 18 years (n=180) meeting the inclusion/exclusion criteria.
7. Randomization and treatment: Patients should receive a 24-hour ambulatory blood pressure monitoring measurement before randomization. After stratification by centers, eligible patients will be randomly divided into two groups, taking losartan 100 mg/hydrochlorothiazide 25 mg fixed combination once a day or amlodipine besylate tablets (5 mg/tablet) + hydrochlorothiazide tablets (25 mg/tablet) once a day.
8. Follow up: 8 weeks.
9. Sample size: a total of 180 patients should be enrolled in the combination.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in September 2018, recruitment will start. Patients enrollment will be performed between October 2018 to August 2024. All patients should be followed up before August 2024.

DETAILED DESCRIPTION:
1. Study name: Efficacy and safety of a single-pill fixed combination of sufficient losartan/hydrochlorothiazide in Chinese hypertensive patients (FOCUS)
2. Medicine: Losartan 100 mg/hydrochlorothiazide 25 mg single-pill fixed combination; amlodipine besylate tablet (5 mg/tablet); hydrochlorothiazide tablets (25 mg/tablet)
3. Rationale: Angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) combined with thiazide diuretic (DIU), which is the preferred combination for most hypertension guidelines. However, the efficacy and safety of losartan 100 mg/hydrochlorothiazide 25 mg single-pill fixed combination evaluated by ambulatory blood pressure are still lack of clinical evidence, especially randomized controlled clinical trials with ambulatory or home blood pressure monitoring as the main evaluation method.
4. Objective The primary objective is to evaluate the efficacy and safety of losartan 100 mg/hydrochlorothiazide 25 mg fixed combination for ambulatory blood pressure after 8 weeks therapy in patients over 18 years with grade 1 or 2 hypertension either newly diagnosed or with blood pressure not controlled with monotherapy. The secondary objective are to compare the 24-hour, daytime, night-time, home and office systolic and diastolic blood pressure between the losartan 100 mg/hydrochlorothiazide 25 mg group and the amlodipine besylate 5 mg/hydrochlorothiazide 25 mg group after 8 weeks of antihypertensive treatment; to compare the changes in blood glucose, blood lipids, blood electrolytes, serum creatinine, blood uric acid and other biochemical parameters.
5. Study design: This study is a multi-center, randomized and controlled clinical trial with two equally sized treatment groups: losartan 100 mg/hydrochlorothiazide 25 mg single-pill combination group and amlodipine besylate 5 mg+hydrochlorothiazide 25 mg group.
6. Study population: Men or Women aged over 18 years (n=180) will be screened, who should never take antihypertensive drugs or stop antihypertensive drugs for more than 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg or who is on monotherapy for at least 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg will be screened. Before randomization, two visits should be performed and 6 clinic blood pressures should be recorded. The average of the 6 clinic blood pressures should be 140-179 mmHg in systolic and/or 90-109 mmHg in diastolic. Regardless of whether the office blood pressure meets the enrollment conditions, a one-week home blood pressure measurement should be performed before randomization. Patient should sign the written consent form before screening and be able to go to the clinic by him/herself. Exclusion criteria included: suspected or confirmed secondary hypertension; history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia; taking other drugs that might affect blood pressure; liver dysfunction, serum creatinine ≥1.5 mg/dL (133 μmol/L), urine protein positive; serum potassium >5.5 mmol/L or <3.5 mmol/L; history of gout or serum uric acid ≥420 μmol/L for man and ≥360 μmol/L for women; elderly care patients; or patients who are participating in other clinical trials.
7. Randomization and treatment: Patients should receive a 24-hour ambulatory blood pressure monitoring measurement before randomization. After stratification by centers, eligible patients will be randomly divided into two groups, taking losartan 100 mg/hydrochlorothiazide 25 mg fixed combination once a day or amlodipine besylate tablets (5 mg/tablet) + hydrochlorothiazide tablets (25 mg/tablet) once a day.
8. Follow up: Sitting office blood pressures should measured by an OMRON device. Medical history should be recorded. Clinical examinations including ambulatory blood pressure, home blood pressure, electrocardiogram, blood and urine routine tests and biochemical tests should be performed. During the 4-week follow-up visit, office blood pressures, serum electrolyte should be measure, adverse events and medication assignment should be recorded. A one-week home blood pressure measurements should be performed immediately before the follow-up visit. During the 8-week follow-up visit, clinical examinations similar with baseline including ambulatory blood pressure, home blood pressure, electrocardiogram, blood and urine routine tests and biochemical tests should be performed.
9. Sample size and statistical analysis: At least 90 eligible patients should be enrolled in each group, and a total of 180 patients should be enrolled in total. Data will be analyzed by using the SAS software. T-tests will be used to compare the parameters between groups and the difference between the two groups with the calculation of 95% confidence interval. In addition, a covariance analysis will also be used in the analysis of baseline parameters.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in September 2018, recruitment will start. Patients enrollment will be performed between October 2018 to August 2024. All patients should be followed up before August 2024. Database construction and statistical analysis will be conducted at the same time, appropriate domestic and international conferences will be selected to publish the research results. The main results will be published in international professional medical journals.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women aged between 18 years will be screened, who should never take antihypertensive drugs or stop antihypertensive drugs for more than 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg or who is on monotherapy for at least 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg will be screened. Before randomization, two visits should be performed and 6 clinic blood pressures should be recorded. The average of the 6 clinic blood pressures should be 140-179 mmHg in systolic and/or 90-109 mmHg in diastolic. Regardless of whether the office blood pressure meets the enrollment conditions, a one-week home blood pressure measurement should be performed before randomization. Patient should sign the written consent form before screening and be able to go to the clinic by him/herself.

Exclusion Criteria:

* suspected or confirmed secondary hypertension; history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia; taking other drugs that might affect blood pressure; liver dysfunction, serum creatinine ≥1.5 mg/dL (133 μmol/L), urine protein positive; serum potassium >5.5 mmol/L or <3.5 mmol/L; history of gout or serum uric acid ≥420 μmol/L for man and ≥360 μmol/L for women; elderly care patients; or patients who are participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 8 weeks
  Number of participants with treatment-related adverse events at the end of 8 weeks of follow-up
Blood pressure control rate | 8 weeks
  The blood pressure controlled rate after 8 weeks of treatment

SECONDARY OUTCOMES:
Ambulatory blood pressure change | 8 weeks
  The changes of ambulatory blood pressure between two treatment groups after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China